CLINICAL TRIAL: NCT02192450
Title: The Effect of Insulin Degludec on Risk of Symptomatic Nocturnal Hypoglycaemia in Subjects With Type 1 Diabetes and High Risk of Nocturnal Severe Hypoglycaemia
Brief Title: Insulin Degludec and Symptomatic Nocturnal Hypoglycaemia
Acronym: HypoDeg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Hvidovre University Hospital (Other); Copenhagen University Hospital, Denmark (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HypoDeg
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Type 1 Diabetes Mellitus; Nocturnal Hypoglycemia; Recurrent Severe Hypoglycaemia
Keywords: Diabetes Mellitus; Hypoglycaemia; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Insulin; Hypoglycaemic Agents; Physiological Effetcs of Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Insulin Resistance | interventions — Insulin Aspart; Insulin Glargine; insulin degludec, insulin aspart drug combination; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin glargine (Active Comparator): Each treatment arm last for 12 months - 3 months of run-in/cross-over and 9 months of maintenance.
  Patients will be randomised (1:1) to treatment with basal-bolus therapy with insulin aspart/degludec or insulin aspart/glargine in random order.
  After 12 months of treatment patients will cross-over to the other basal-bolus therapy.
  Insulin degludec and insulin glargine is administered once daily at the evening meal and insulin aspart is administered three times daily before the main meals.
  Interventions: Drug: Insulin aspart/glargine
- Insulin degludec (Experimental): Each treatment arm last for 12 months - 3 months of run-in/cross-over and 9 months of maintenance.
  Patients will be randomised (1:1) to treatment with basal-bolus therapy with insulin aspart/degludec or insulin aspart/glargine in random order.
  After 12 months of treatment patients will cross-over to the other basal-bolus therapy.
  Insulin degludec and insulin glargine is administered once daily at the evening meal and insulin aspart is administered three times daily before the main meals.
  Interventions: Drug: Insulin aspart/degludec

INTERVENTIONS:
Drug: Insulin aspart/glargine
  Other Names: NovoRapid; Lantus
  Arms: Insulin glargine
Drug: Insulin aspart/degludec
  Other Names: NovoRapid; Tresiba
  Arms: Insulin degludec

SUMMARY:
The purpose of this study is to determine whether insulin degludec compared to insulin glargine can reduce the risk of symptomatic nocturnal hypoglycaemia in subjects with the greatest potential benefit from optimised insulin treatment, which are patients with type 1 diabetes and high risk of nocturnal severe hypoglycaemia.

DETAILED DESCRIPTION:
Background: Insulin degludec is a novel insulin analogue that may reduce the risk of mild nocturnal hypoglycaemia in type 1 diabetes. Patients with type 1 diabetes and recurrent severe hypoglycaemia (high risk patients) are also burdened by nocturnal hyoglycaemia (mild and silent). These episodes may contribute to the developement of hormonal counterregulatory failure and hypoglycaemia unawareness, which in turn increases the risk of further hypoglycaemic episodes, especially epiosdes of severe hypoglycaemia.The effect of insulin degludec on risk of mild nocturnal hypoglycaemia in subjects with type 1 diabetes and high risk of severe hypoglycaemia compared to insulin glargine is to be investigated.

Study design and intervention: A controlled, cross-over multi-centre study in a Prospective, Randomised, Open, Blinded Endpoint (PROBE) design. Each treatment period last for 12 months. Patients will be randomised to treatment with basal-bolus therapy with insulin aspart/degludec or insulin aspart/glargine in random order. Endpoints will be assessed during the last 9 months of each treatment arm.

Subjects: 175 type 1 diabetic patients with a history of one or more episodes of nocturnal severe hypoglycaemia during the proceeding two years.

Method: Patients will record all events of symptomatic (mild), asymptomatic (silent) and severe hypoglycaemia in a diary. All events of symptomatic nocturnal and severe hypoglycaemia must also be reported by telephone within 24 hours. Patients will be instructed to do and record self-monitored blood glucose (SMBG) i.e. 4-point profiles twice per week (blood glucose before breakfast, before lunch, before dinner and before bedtime).

Outcomes: See "Outcome Measures". Concerning the primary endpoint all possible symptomatic nocturnal hypoglycaemic episodes will be adjudicated by an independent endpoint committee consisting of diabetes specialists blinded to the individual patient insulin regimen.

Safety: Adverse reactions

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes > 5 years
* One or more episodes of nocturnal severe hypoglycaemia during the preceding two years
* Treated with multiple dose insulin injection (>2) or insulin pump. Both human insulin and insulin analogues are allowed
* Willingness to a once daily (OD) regimen concerning insulin degludec and insulin glargine
* Willingness to do self-monitoring of blood glucose (SMBG) and keep a diary
* Signed informed consent

Exclusion Criteria:

* History of primary and secondary adrenal insufficiency, growth hormone deficiency, or untreated myxoedema
* History of unstable angina or major cardiovascular events (myocardial infarction, coronary re-vascularisation, transient ischaemic attack, or stroke within the last three months)
* Heart failure, New York Heart Association (NYHA) class IV
* History of malignancy unless a disease-free period exceeding five years
* History of alcohol or drug abuse
* Treatment with glucose lowering agent(s) other than insulin
* Pregnant or lactating women
* Women of childbearing potential who are not using chemical (P-pills or gestagen depots) or mechanical (intra-uterine device) contraception
* Participation in another investigational drug study within the last 3 months
* Inability to understand the informed consent
* HbA1c > 86 mmol/mol (10%)
* Shifting working hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-01; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Symptomatic nocturnal hypoglycaemia | 9 months (3-12) of each treatment period

SECONDARY OUTCOMES:
Severe hypoglycaemia (total, night-time, daytime) | 9 months (3-12) of each treatment period
Any nocturnal hypoglycaemia (incl. asymptomatic/silent events) | 9 months (3-12) of each treatment period
Any daytime hypoglycaemia (symptomatic, asymptomatic/silent and severe) | 9 months (3-12) of each treatment period
Any CGM recorded hypoglycaemia (symptomatic, asymptomatic/silent and severe) | 2 x 6 days in each treatment arm
Any in-hospital nocturnal hypoglycaemia (incl. asymptomatic/silent events) | 2 overnight stays in each treatment arm
Change in HbA1c | From baseline to after 12 months of treatment
Change in glycaemic variability | 4 x overnight stays and 4 x 6 days of CGM
Insulin doses | End of each treatment period
Quality of life incl. pre-depression scale | At baseline, cross-over and after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Pedersen-Bjergaard, MD, DMSc, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hilleroed, Denmark

REFERENCES:
- [Derived] Brosen JMB, Agesen RM, Alibegovic AC, Ullits Andersen H, Beck-Nielsen H, Gustenhoff P, Krarup Hansen T, Hedetoft CGR, Jensen TJ, Stolberg CR, Bogh Juhl C, Lerche SS, Norgaard K, Parving HH, Tarnow L, Thorsteinsson B, Pedersen-Bjergaard U. Continuous Glucose Monitoring-Recorded Hypoglycemia with Insulin Degludec or Insulin Glargine U100 in People with Type 1 Diabetes Prone to Nocturnal Severe Hypoglycemia. Diabetes Technol Ther. 2022 Sep;24(9):643-654. doi: 10.1089/dia.2021.0567. Epub 2022 Jun 22. PMID 35467938
- [Derived] Agesen RM, Alibegovic AC, Andersen HU, Beck-Nielsen H, Gustenhoff P, Hansen TK, Hedetoft C, Jensen T, Juhl CB, Lerche SS, Norgaard K, Parving HH, Tarnow L, Thorsteinsson B, Pedersen-Bjergaard U. The effect of insulin degludec on risk of symptomatic nocturnal hypoglycaemia in adults with type 1 diabetes and high risk of nocturnal severe hypoglycaemia (the HypoDeg trial): study rationale and design. BMC Endocr Disord. 2019 Jul 23;19(1):78. doi: 10.1186/s12902-019-0408-x. PMID 31337371